CLINICAL TRIAL: NCT07015619
Title: Effects of Task Specific Balance Training VS Task-oriented Basketball Training on Balance and Motor Skills in Children With Developmental Delay
Brief Title: Task Specific vs Basketball-Based Balance Training in Children With Developmental Delay
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shalamar Institute of Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: ShalamarSSAHS
Record Dates: First submitted 2025-06-03; First posted 2025-06-11 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Development Delay
Keywords: DD; TSBT; TOBT
MeSH Terms: conditions — Learning Disabilities

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Task Specific Balance Training (Other): Group A: Participants will perform Task specific balance training. The interventions will be performed three times per week, for total of 24 sessions, within 8 weeks. There will be a Warm-up session of 5 minutes that will include active exercises such as ankle pumps and arm swings. Sufficient rest intervals during each training session. In each session, participants will perform three repetitions of each exercise. For static balance, the exercises will include one-leg standing, tandem standing, heel-to-toe walking, and stride sitting on a peanut ball. For dynamic balance, the exercises will include stepping over obstacles, walking on a balance beam, side-stepping, and walking in a straight line while balancing a ball on a board
  Interventions: Other: Task Specific Balance Training
- Task-oriented Basketball Training (Other): Group B: Participants will perform Task oriented basketball training. The interventions will be performed three times per week, for total of 24 sessions, within 8 weeks. There will be warm up session of 5 minutes that will include active exercises that are ankle pumps and arm swing. Sufficient rest interval during each training session. In one session, participants will perform three repetitions for each exercise. Exercises are basic dribbling, passing and catching, partner based passing and catching, target shooting, hurdle jumping, wall catching, skipping hoops and cone drills.
  Interventions: Other: Task-oriented Basketball Training

INTERVENTIONS:
Other: Task Specific Balance Training — Group A participants will undergo Task Specific Balance Training. It is a rehabilitation approach that focus on improving balance by practicing specific balance related tasks.
  Arms: Task Specific Balance Training
Other: Task-oriented Basketball Training — Group B participants will undergo Task-oriented Basketball Training. It is a rehabilitation approach that focuses on balance, coordination and gross motor skills through specific basketball related tasks.
  Arms: Task-oriented Basketball Training

SUMMARY:
To compare the effects of task specific balance training vs task-oriented basketball training on balance and motor skills in children with developmental delay

DETAILED DESCRIPTION:
Developmental delay (DD) in children presents as delays in motor, cognitive, and social skills that are essential for daily life. The most affected areas are gross motor and balance abilities. These are crucial for mobility, independence, and participation in physical activities. Physiologically, gross motor function involves the coordinated work of the neuromuscular system, proprioceptive input, and cerebellar processing. These systems help maintain balance and perform postural transitions. When delayed, they can lead to poor coordination, postural instability, and reduced physical activity.

Globally, developmental delay affects an estimated 5% to 15% of children. The rate is higher in low- and middle-income countries due to malnutrition, prenatal issues, and lack of early intervention. In Pakistan, 37.9% of children in a Karachi-based study had developmental delay. The condition was more common in slum areas.

Task-specific balance training (TSBT) aims to improve sensory integration and postural control. It uses targeted tasks that challenge balance in static and dynamic situations. A randomized trial showed significant improvements in sensory organization and balance in children with developmental disorder who received TSBT. Task-oriented basketball training (TOBT), on the other hand, combines cognitive and motor challenges. It uses sport-specific activities to enhance balance, coordination, and fitness. Research shows that TOBT improves motor skill-related fitness in children with DD. Previous research has found that both task-specific balance training and task-oriented basketball training independently help children with developmental delay by improving their balance and movement skills. However, no studies have directly compared these two methods to see which one works better. This study will do that comparison. The results will help therapists choose the best training approach for these children, improving rehabilitation strategies.

This study signifies the importance of effects of Task Specific Balance Training and Task-oriented Basketball Training in enhancing balance and motor skills in developmentally delayed children which ultimately contributes towards making them a functional independent individual of our community. Improved balance and coordination may enhance children active participation in community activities, reducing caregiver dependence. This study will contribute optimizing rehabilitation strategies for pediatric population with motor and balance impairments.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 5-12

  * Diagnosed with DD
  * Able to follow instruction
  * Male and female are included

Exclusion Criteria:

* • Neurological conditions other than DD

  * Musculoskeletal deformities
  * Visual or hearing impairments
  * Participants who are unable to engage in the assigned interventions due to physical or cognitive limitations

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2025-06-28 (Estimated); Primary Completion 2025-10-29 (Estimated); Study Completion 2025-11-29 (Estimated)

PRIMARY OUTCOMES:
Improved balance | 8 WEEKS
  Pediatric Balance Scale (PBS) is a 14 item performance based measure, assessing balance in sitting, standing and during functional tasks. Each item is scored on a scale of 0-4, with higher scores indicating better balance

SECONDARY OUTCOMES:
Improved motor skills | 8 WEEKS
  Gross Motor Function Measure (GMFM-88) is a standardized observational tool, measuring gross motor function in five domains: lying/rolling(17 items), sitting(20 items), crawling/kneeling(14 items), standing(13 items) and walking/running/jumping(24 items). The score for each dimension is presented as the percentage of maximum score for the dimension. Each of 88 items is scored on a 4-point ordinal scale(0 = does not initiate, 1 = initiates, 2 = partially completes, 3 = completes). Minimum possible total score is 0% and maximum possible score score is 100%. Higher scores represent better gross motor function and improvement.